CLINICAL TRIAL: NCT01347957
Title: Safety and Efficacy of Nitric Oxide Gel in Promoting Hair Growth in Male Human Subjects With Androgenetic Alopecia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR98-IRB-231
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Alopecia Androgenica
MeSH Terms: interventions — Nitric Oxide; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitric Oxide (NO) Gel (Experimental)
  Interventions: Other: Nitric Oxide (NO) Gel
- Placebo Gel (Placebo Comparator)
  Interventions: Other: Placebo gel

INTERVENTIONS:
Other: Nitric Oxide (NO) Gel — Nitric Oxide (NO) Gel is created by premixing of contents from 2 separate gel bottles. The first bottle, NO gel, is a solution of sodium nitrite (14.6mM) in distilled water with hydroxyethylcellulose (molecular weight 50,000-1,250,000) added for gel formation. The second bottle, Releasing-stimulator gel, is a solution of maleic acid (14.6mM) and ascorbic acid (14.6mM) in distilled water with hydroxyethylcellulose added for gel formation.
  Arms: Nitric Oxide (NO) Gel
Other: Placebo gel — The placebo gel is created by premixing of contents from 2 separate gel bottles. The first bottle is phosphate-buffered saline. The second bottle is the second gel bottle (Releasing-stimulator gel) as described in experimental arm.
  Arms: Placebo Gel

SUMMARY:
Preclinical studies showed the Nitric Oxide (NO) gel significantly promoted hair follicle formation and growth in both rat and mouse models. The NO gel induced major physiological, developmental, and structural changes in the skin of mammals to increase the number of hair follicles, follicle stem cell development and regeneration as well as hair shaft elongation, and accelerated hair growth rate. Based on our animal model findings, the investigators hypothesize that the nitric oxide releasing gel could be used as a medical treatment for hair growth in humans. The objective of this trial is to evaluate the safety and efficacy of this NO gel (XN-001), in comparison with a placebo gel in subjects in a 24-week treatment schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects >= 20 and <= 65 years of age.
2. Subjects with hair loss caused by androgenetic alopecia.
3. Subjects who are healthy without any serious diseases that require hospitalization during the study period.
4. Subjects who are capable of understanding and having signed the Informed Consent Form after detailed description of the treatment procedures and potential risks and benefits.

Exclusion Criteria:

1. Subjects who received any treatment for hair loss within 6 months or finasteride within 12 months
2. Subjects with diagnosis of cancer and is still on active therapies.
3. Subjects with diagnosis of an active disease and is still under regular treatment for this disease
4. Subjects with hair loss caused by a known chronic disease.
5. Subjects who are on vasodilators or other medication with pharmacological actions that may lead to excessive formation of nitric oxide or may accentuate drug effects due to excessive formation of nitric oxide.
6. Subjects with thyroid disease.
7. Subjects iron-deficiency anemia.
8. Subjects with skin diseases of the scalp, including severe seborrhoeic dermatitis, psoriasis, lichenoid eruption, tinea capitis, or other scalp infections or infestations
9. Subjects with any known allergic reaction to any ingredient in the 2 gel preparations.
10. Subjects who have been enrolled into any clinical study in the preceding 6 months prior to randomization.
11. Subjects who have taken medications that are known to induce hypotrichosis or hypertrichosis.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the difference in TAHC between baseline and after 24-week treatment (NO vs. placebo groups). | 24 weeks

SECONDARY OUTCOMES:
The secondary efficacy end point will be subjective assessment of improvement. | 24 weeks
  Subjects will be instructed to fill out a questionnaire at week 24 to evaluate the overall condition of hair loss in comparison with baseline.
  Subjects will be evaluated for any possible adverse effects of study drug and any symptoms and signs of scalp irritation (stinging, burning, itching)

CONTACTS AND LOCATIONS:
Overall Officials: Chih JUNG HSU, Principal Investigator — Dermatological department, CMUH
Locations (1):
- Dermatological Department, CMUH, Taichung, Taiwan